CLINICAL TRIAL: NCT02187107
Title: An Open Label Trial of TMC114/Rtv in HIV-1 Infected Subjects Who Were Randomized in the Trials TMC114-C201, TMC114-C207 or in Sponsor Selected Phase I Trials
Brief Title: A Study to Assess the Long-term Safety and Tolerability of TMC114/Rtv in HIV-1 Infected Participants After Rolling-over From Other TMC114 Trials
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005848; TMC114-C208 (Other: Tibotec Pharmaceuticals Limited, Ireland)
Record Dates: First submitted 2014-02-25; First posted 2014-07-10 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: HIV
Keywords: HIV; AIDS; TMC114; Ritonavir; Norvir; Darunavir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC114 + rtv (Experimental): Every participant recieves 2 tablets of TMC114, 300 mg, combined with one tablet of rtv (ritonavir), 100mg, orally twice daily, every 12 hours
  Interventions: Drug: TMC114; Drug: rtv

INTERVENTIONS:
Drug: TMC114 — 300 mg tablets of TMC114 ethanolate with microcrystalline cellulose, colloidal silicon dioxide, crospovidone, magnesium stearate, and Opadry® Orange
Drug: rtv — 100 mg tablet of Norvir®
  Other Names: Norvir

SUMMARY:
The purpose of this study was primarily to assess the long-term safety and tolerability of TMC114/rtv in addition to an individually optimized background antiretroviral therapy in HIV-1 infected participants. In addition, antiviral activity and immunological effect were also evaluated.

DETAILED DESCRIPTION:
This was a phase II, open label, multicenter trial of an investigational protease inhibitor TMC114 in the presence of ritonavir (rtv) in HIV-1 infected participants who were randomized in trials TMC114-C201, TMC114-C207 or in sponsor selected phase I trials and who might derive benefit from TMC114 therapy, as judged by the investigator.

The trial consisted of a screening period of a maximum of 4 weeks, a 96-week treatment period and a 4-week follow-up period. The maximal trial duration for each participant was104 weeks. During the treatment period, all participants were receiving TMC114 in combination with RTV, orally, as 600/100 mg dose twice daily, in addition to an individually optimized background regimen of antiretroviral (ARV) therapy, selected by the investigator at a baseline of the study.

Sponsor provided a follow-up treatment with TMC114 for all participants who continued to benefit from treatment with TMC114/RTV until it became commercially available for the participant. Participants, who completed the 96 weeks of treatment period with TMC114, had the opportunity to roll over to the extension of this trial, if TMC114 was not locally commercially available.

ELIGIBILITY:
Inclusion Criteria

* Must be diagnosed with HIV
* Previously randomized in trials TMC114-C201, TMC114-C207 or in sponsor selected Phase I trials
* Agreed to take at least 2 antiretroviral agents from baseline onwards
* Could comply with the protocol requirements
* General medical condition, in the investigator's opinion, was not interfering with the assessments and the conduct of the trial

Exclusion Criteria:

* A disallowed concomitant therapy
* Current or past history of active alcohol and/or drug use
* Pregnant or breast-feeding females
* Any active or unstable medical condition (e.g., tuberculosis; cardiac dysfunction; pancreatitis; acute viral infections)
* Clinical or laboratory evidence of active liver disease, liver impairment/dysfunction or cirrhosis
* Clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication
* Laboratory abnormalities at screening (criteria variable according to the test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-01; Primary Completion 2005-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of TMC114/RTV 600/100 mg combination | Baseline, up to the end of follow-up period (approximatelly 100 weeks)

SECONDARY OUTCOMES:
Number of patients with HIV-1 plasma viral load level <50 copies/mL (TLOVR, non-VF censored) | Week 48, Week 96
  The Time to Loss of Virologic Response (TLOVR) algorithm will be used to derive response. Response will be confirmed at 2 consecutive visits and participants who discontinue will be considered nonresponders after discontinuation. Resuppression after confirmed virologic failure will be considered as failure. Virologic Failure will include participants who are rebounders (ie, confirmed viral load >= 50 copies/mL after being a responder) or who were never suppressed (no confirmed viral load <50 copies/mL); non-VF censored: participants who discontinue treatment due to reason other than Virologic Failure will be excluded.
Change in CD4 cells absolute count | Week 48, Week 96
  The immunologic change will be determined by changes in absolute values for CD4 cells.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (11):
- Darlinghurst, Australia
- Vienna, Austria
- Ghent, Belgium
- Copenhagen, Denmark
- Germany (4):
  - Berlin
  - Hamburg
  - Hanover
  - Munich
- Szczecin, Poland
- Saint Petersburg, Russia
- London, United Kingdom

REFERENCES:
- See also: An Open Label Trial of TMC114/Rtv in HIV-1 Infected Subjects Who Were Randomized in the Trials TMC114-C201, TMC114-C207 or in Sponsor Selected Phase I Trials — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1455&filename=CR005848_CSR.pdf